CLINICAL TRIAL: NCT03096210
Title: Comparison of the Clinic, Radiographic and Histological Effects of Allograft and T-PRF (Titanium-Prepared Platelet Rich Fibrin) Materials in the Sinus Lifting Procedure. Preliminary Results From a Pilot Randomised Controlled Trial
Brief Title: Titanium-Prepared Platelet Rich Fibrin in the Sinus Lifting Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ebru Olgun Erdemir, Prof.Dr., Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/05
Record Dates: First submitted 2017-03-08; First posted 2017-03-30 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Maxillary Sinus
Keywords: Maxillar sinus; Titanium-Prepared Platelet Rich Fibrin; Allograft; implant
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium-Prepared Platelet Rich Fibrin (Other): After careful elevation of the schneiderian membrane without perforation,T-PRFs were only used in the test group.
  Interventions: Other: Titanium-Prepared Platelet Rich Fibrin
- Allograft (CTBA Allograft) (Other): After careful elevation of the schneiderian membrane without perforation, allograft was only used for augmentation of the sinus floor in the control group.
  Interventions: Other: Allograft (CTBA Allograft)

INTERVENTIONS:
Other: Titanium-Prepared Platelet Rich Fibrin — Blood samples were collected from the each participant's arm in the test group by 20 ml syringe and then was transferred into 10ml grade IV titanium tube without anticoagulant. After centrifugation of blood samples (2800 rpm, 12 minutes) at room temperature, the T-PRF clot was removed from the tubes with sterile tweezers. 6 blood tubes were collected for a sinus floor elevation/lifting operation and 6 T-PRFs were prepared for each participant.
  Arms: Titanium-Prepared Platelet Rich Fibrin
Other: Allograft (CTBA Allograft) — After careful elevation of the schneiderian membrane without perforation, allograft was only used for augmentation of the sinus floor in the control group.
  Arms: Allograft (CTBA Allograft)

SUMMARY:
This study evaluates the radiographic, histological and clinical comparisons of the completely autologous T-PRF or allograft effectiveness at the maxillary sinus elevation procedure.

DETAILED DESCRIPTION:
Participants randomly divided into 2 groups and the test group had a Schneiderian membrane elevation with using balloon lifting technique and after that sinus was filled with T-PRF produced from the patients' blood and 4 months waiting period has been entered. At the end of the 4th month, the bone samples were received from the implant slots and sent to histological evaluation. After 3 months, implant stability was measured and recorded. In the control group, the same procedures were followed and sinus was filled with only allograft. Waiting period was changed to 6 months for this group.

ELIGIBILITY:
Inclusion Criteria:

* Participants having been diagnosed to display a residual crest height of less than 5mm in posterior maxilla and non-smokers were included.

Exclusion Criteria:

* Participants with blood platelet disorders, infectious and metabolic diseases, ongoing chemotherapy or radiotherapy, history of chronic sinusitis associated with maxillary sinuses, taking any antibiotics and/or anti-inflammatory drugs were excluded.

Ages: 42 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03-11 (Actual); Primary Completion 2014-11-28 (Actual); Study Completion 2015-03-02 (Actual)

PRIMARY OUTCOMES:
Histological Examination | At the first 4 and 6th months post surgery for the test and control groups, respectively.
  Percentage (%) of new and old trabeculae formation post surgery

SECONDARY OUTCOMES:
Radiological Examination | Within the first 4 and 6 months
  Density (hu) measurements
Implant stability measurements | Within the 3 months after implant surgery
  Implant Stability Quotient values (50-80 ISQ)

IPD SHARING:
Plan to Share IPD: No